CLINICAL TRIAL: NCT05147896
Title: Semaglutide Anti-Atherosclerotic Mechanisms of Action Study in Type 2 Diabetes Patients
Acronym: SAMAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrej Janez, MD, PhD, Prof, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMCLjubljana20210043
Record Dates: First submitted 2021-11-21; First posted 2021-12-07 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; Atherosclerosis
Keywords: semaglutide; atherosclerosis; diabetes mellitus type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Arm (Active Comparator): Beside metformin and sulphonyl urea treatment, the active, interventional arm, will be receiving Semaglutide Oral Tablets as per protocol, 3 mg for the first month, 7 mg in the second month and 14 mg form the third month onwards.
  Interventions: Drug: Semaglutide Oral Tablet
- Comparative Arm (No Intervention): This group will not be receiving the additional therapy besides metformin and sulphonyl urea treatment. After 6 months a revaluation of glycemic control will be performed, if needed, rescue therapy with basal insulin will be implemented.

INTERVENTIONS:
Drug: Semaglutide Oral Tablet — Semaglutide Oral Tablets will be introduced to the active arm as per protocol for regular therapy introduction.
  Other Names: Rybelsus
  Arms: Interventional Arm

SUMMARY:
Diabetes is a chronic disease characterized by chronic hyperglycaemia, causing microvascular and macrovascular complications. The latter lead to various disabilities: blindness, end-stage renal failure, nerve damage, formation of leg ulcers, and atherosclerosis. In people with type 2 diabetes, the probability of these atherosclerosis associated complications is twice as high as in people without diabetes. Cardiovascular diseases are also the main cause of mortality in people with diabetes.

Preventive measures are therefore crucial. In people with type 2 diabetes, in addition to good glycaemic control, the choice of antidiabetic drugs is also important. Large-scale research has shown that certain glucagon-like peptide (GLP-1) receptor agonists, in addition to improving the regulation of diabetes, also have a significant effect on reducing the macrovascular complications. It is now possible to use semaglutide, a GLP-1 receptor agonist, in the tablet form. Semaglutide lowers blood sugar only when the blood sugar value rises, due to food in the digestive tract, Thus, not increasing the risk of hypoglycaemia. In addition, semaglutide has a significant effect on weight loss and very beneficial, protective effects on the cardiovascular system. Large studies have shown that in its injectable form, it significantly reduces the incidence of cardiovascular death in patients with type 2 diabetes.

Therefore, the aim of the present study is to examine how semaglutide provides protective effects on the cardiovascular system and reduces the risk of diabetes type 2 associated complications.

The present study will include 100 people with type 2 diabetes and last for 12 months. The subjects will receive a semaglutide oral tablet daily in addition to their current treatment (combination of metformin and a sulphonyl urea). At the beginning of the study, after 6 months and at the end of the study (after 12 months of treatment), a detailed clinical examination will be performed and blood will be taken for laboratory parameters. In addition to basic blood tests, inflammatory and oxidative stress parameters, as well as lipid fractions parameters will also be assessed. Ultrasound examination of the changes in the carotid arteries and measures of additional properties of the arteries will also be performed. The confidentiality of the data of the participants in the research will be ensured, as the data obtained during the investigation will be encrypted before processing.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* therapy including at least metformin 1000 mg and sulphonyl urea at least half of the maximal dose
* BMI > or = 30 kg/m2
* HbA1c < or = 8,5%
* associated risk factors including smoking, dyslipidaemia, arterial hypertension, chronic kidney disease stage 1 to 3.

Exclusion Criteria:

* therapy with injectable GLP-1 receptor agonist ongoing or was taking place in the last year
* manifested cardiovascular disease
* heart failure
* chronic kidney disease stages 4 and 5
* advanced liver disease
* proliferative retinopathy or maculopathy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in morphological arterial wall characteristics | 1 year
  Ultrasonographic assessment of cIMT (in millimetres)
Change in functional arterial wall characteristics | 1 year
  Endothelial function assessment by EndoPAT
Change in structural arterial wall characteristics | 1 year
  Arterial stiffness assessment by Sphygmocor device (in meters per second)

SECONDARY OUTCOMES:
Change in atherogenic small dense low-density lipoproteins (sdLDL) | 1 year
  Assessment by gel electrophoresis
Change in glycated haemoglobin (HbA1c) | 1 year
  Assessment by biochemical methods
Change in high sensitivity C-reactive protein (hsCRP) | 1 year
  Assessment by biochemical methods
Correlations between changes in rate of cIMT reduction, % of endothelial function improvement and rate of arterial stiffness reduction on one hand and changes in concentration of sdLDL, % of HbA1c and concentration of hsCRP on the other | 1 year
  Statistical methods

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janež, Prof, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- UMC Ljubljana, Diabetes Outpatient Clinic, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janic M, Rizzo M, Cosentino F, Pantea Stoian A, Lunder M, Sabovic M, Janez A. Effect of Oral Semaglutide on Cardiovascular Parameters and Their Mechanisms in Patients with Type 2 Diabetes: Rationale and Design of the Semaglutide Anti-Atherosclerotic Mechanisms of Action Study (SAMAS). Diabetes Ther. 2022 Apr;13(4):795-810. doi: 10.1007/s13300-022-01226-y. Epub 2022 Mar 8. PMID 35258841